CLINICAL TRIAL: NCT03603379
Title: A Pharmacokinetic Phase 1 Study of Anti-epidermal Growth Factor Receptor (EGFR) -Immunoliposomes Loaded With Doxorubicin in Patients With Relapsed or Refractory High-grade Gliomas
Brief Title: Doxorubicin-loaded Anti-EGFR-immunoliposomes (C225-ILs-dox) in High-grade Gliomas
Acronym: GBM-LIPO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-01160; me17Kasenda2
Record Dates: First submitted 2018-07-17; First posted 2018-07-27 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Glioblastoma
Keywords: anti- EGFR- immunoliposomes
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- C225-ILs-dox i.v. (Experimental): C225-ILs-dox administered intravenously
  Interventions: Drug: C225-ILs-dox

INTERVENTIONS:
Drug: C225-ILs-dox — C225-ILs-dox will be administered at a dose of 50 mg/m2. i.v., on day 1 of each cycle, cycle length is 28 days. In total, 4 cycles are planned to be applied.

SUMMARY:
Anti-EGFR-immunoliposomes loaded with doxorubicin (C225-ILs-dox) are given intravenously in patients with relapsed or refractory high-grade gliomas.

The pharmacokinetics of C225-ILs-dox in peripheral blood (PB), cerebro-spinal fluid (CSF) and resected tumour tissue will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent according to International Conference on Harmonization (ICH)/Good Clinical Practice (GCP) regulations before registration and prior to any trial specific procedures
2. Patients with relapsed histologically proven glioblastoma ≥ 18 years of age.
3. Patients need to have at least one line of treatment with combined radio-chemotherapy
4. EGFR amplification. EGFR amplification will be tested by comparative genomic hybridization (CGH) method. EGFR will be considered amplified if the value is 0.15 above the average signal of chromosome 7.
5. Evaluable disease on MRI brain scan
6. Adequate bone marrow function: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L
7. Adequate hepatic function: bilirubin ≤ 1.5 x upper limit of normal (ULN), aspartate aminotransferase (AST), Alanin-Aminotransferase (ALT) and alkaline phosphatase (AP) ≤ 2.5 x ULN
8. Adequate renal function: serum creatinine ≤ 1.5 x ULN and calculated creatinine clearance > 30 mL/min, according to the formula of Cockcroft-Gault
9. Adequate cardiac function: Left ventricular Ejection Fraction (LVEF) ≥ 50% as determined by either echocardiography (ECHO) or radionuclide angiocardiography (MUGA) in addition to pre- (brain-type natriuretic Peptide) BNP from peripheral blood
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (0=Fully active, able to carry on all pre-disease performance without restriction, 1=Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2=Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours).
11. No contraindications for lumbar puncture
12. Women with child-bearing potential have to use effective contraception, are not allowed to be pregnant and have to agree not to become pregnant during trial treatment and during the 6 months thereafter. A negative pregnancy test before inclusion into the trial is required for all women with child-bearing potential.

Exclusion Criteria:

1. History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration except for adequately treated cervical carcinoma in situ and localized non-melanoma skin cancer.
2. Lack to provide written informed consent
3. Previous therapy with more than 240 mg/m2 of doxorubicin or more than 450 mg/m2 of epirubicin
4. Any serious underlying medical condition (at the judgement of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes, etc.)
5. Breastfeeding and pregnancy
6. Participation in any investigational drug trial within 4 weeks preceding treatment start
7. Any concomitant drugs contraindicated when administering Erbitux™ or Caelyx™ according to the Swissmedic-approved product information
8. Known hypersensitivity to trial drug(s) or to any component of the trial drug(s)
9. Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Ratio of C225-ILs-dox concentration | 24 hours after first C225-ILs-dox application
  Ratio of C225-ILs-dox concentration in cerebro-spinal fluid over the C225-ILs-dox concentration in peripheral blood.

SECONDARY OUTCOMES:
Tumour response according to RANO criteria on the final MRI scan | At the end of 4 treatment cycle 4 (each cycle is 28 days)
  Tumour response according to RANO criteria; RANO criteria: divides response into four types of response based on imaging (MRI) and clinical features: complete response partial response stable disease progression
Best achieved tumour response (1st or second MRI scan) during treatment phase according to RANO criteria ( | between day 28 and day 104
  1st or second MRI scan during treatment phase according to RANO criteria. RANO criteria: divides response into four types of response based on imaging (MRI) and clinical features: complete response partial response stable disease progression
Event free survival | 12 months
  Defined as the time between registration to progression, termination of therapy for toxicity, or death whichever occurs first.
Progression free survival | 12 months
  Defined as the time between registration to progression or death whichever occurs first
Overall survival | 12 months
  Defined as the time between registration to death due to any cause
Toxicity as graded by the CTCAE Version 4.0 | 12 months
  CTCAE grade 4 Life-threatening consequences; urgent intervention indicated; Neutrophils < 0.5 x 109/l or Platelets < 25 x 109/l; febrile neutropenia

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Laeubli, MD, Principal Investigator — Dep. Oncology University Hospital Basel
Locations (2):
- Switzerland (2):
  - Kantonsspital Aarau (KSA), Oncology, Aarau
  - Department of Oncology University Hospital Basel, Basel

REFERENCES:
- [Derived] Kasenda B, Konig D, Manni M, Ritschard R, Duthaler U, Bartoszek E, Barenwaldt A, Deuster S, Hutter G, Cordier D, Mariani L, Hench J, Frank S, Krahenbuhl S, Zippelius A, Rochlitz C, Mamot C, Wicki A, Laubli H. Targeting immunoliposomes to EGFR-positive glioblastoma. ESMO Open. 2022 Feb;7(1):100365. doi: 10.1016/j.esmoop.2021.100365. Epub 2022 Jan 5. PMID 34998092